CLINICAL TRIAL: NCT06325514
Title: The Application of an Artificial Intelligence Based Program to Classify Oral Cavity Findings Based on Clinical Image Analysis
Brief Title: Artificial Intelligence Based Program to Classify Oral Cavity Findings Based on Clinical Image Analysis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noran Ayman Mohammad Ismael Abdel-Moaty, Principal Investigator, Cairo University
Other Study IDs: NA2024
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Oral Cancer; Oral Lichen Planus; Fordyce Granule; Leukoplakia; Erythroplakia; Leukoedemas, Oral; Lichenoid Reaction
MeSH Terms: conditions — Mouth Neoplasms; Lichen Planus, Oral; Leukoplakia; Erythroplasia; Leukoedema, Oral; Lichenoid Eruptions

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal/variations of normal anatomical landmarks: patients that have normal oral findings or variations of normal anatomical landmarks such as: leukoedema, fordyce granules, linea alba, physiological pigmentations, torus palatinus, torus mandibularis, geographic tongue, fissured tongue
  Interventions: Diagnostic Test: Artificial intelligence based program
- low risk referral: patients that needs referral for a low risk of malignant transformation disease, such as: hemangiomas, fibromas, oral apthous ulcers, candidal infections, pemphigus valgaris, petechiae, frictional keratosis, smokers' melanosis.
  Interventions: Diagnostic Test: Artificial intelligence based program
- high risk referral: patients that needs referral for a high risk of malignancy or a premalignant disease, such as: oral lichen planus, leukoplakia, erythroplakia, squamous cell carcinoma.
  Interventions: Diagnostic Test: Artificial intelligence based program

INTERVENTIONS:
Diagnostic Test: Artificial intelligence based program — the AI based program is based on image analysis

SUMMARY:
This study aims to develop an AI program that can classify oral findings into Normal/variation of normal or an oral disease by clinical photos analysis, aiding in lowering the percentages of false positive and false negative diagnosis of oral diseases.

DETAILED DESCRIPTION:
Early diagnosis of oral lesions, particularly oral cancer, is crucial for enhancing prognosis, facilitating early intervention and care with the intention of lowering disease-related mortality.

Since conventional oral examination (COE) is the most used method in identifying oral lesions, the average dental practitioner's experience is a decisive factor in early diagnosis.

Visual examination lacks specificity and sensitivity since its highly subjective. Unfortunately, Studies show that the majority of dentists lack expertise in early detection of the disease, resulting in false negative diagnosis of oral lesions.

General practitioners are found to either delay the referral of a suspected oral lesion to an Oral Medicine specialist, or referring numerous false positive cases, unnecessarily pushing the patients into a state of anxiousness and cancer phobia. False positive referrals overburden the specialists, which will eventually cause delayed diagnosis of true positive cases due to the oversaturation with false positive ones.

diagnostic research scope shifts towards noninvasive, easy chair side methods with higher accuracy for early detection of oral lesions. Recent approaches towards using machine based programs indicate that this machine-learning method may be useful in the detection and diagnosis of oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old
* Candidates with normal oral cavity findings
* Candidates with variations of oral cavity findings
* Candidates with different oral lesions

Exclusion Criteria:

• Patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients should be above 18 years old, with no maximum age limit. Normal oral cavity findings, variations of oral anatomical landmarks, patients with oral lesions are all included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
risk stratification | 3 months to develop the program
  patient is either normal with no risk or need for referral, low risk of malignant transformation disease, high risk of malignant transformation disease.

CONTACTS AND LOCATIONS:
Overall Officials: Noran AM AbdelMoaty, MsC, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry, CairoU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khanagar SB, Al-Ehaideb A, Maganur PC, Vishwanathaiah S, Patil S, Baeshen HA, Sarode SC, Bhandi S. Developments, application, and performance of artificial intelligence in dentistry - A systematic review. J Dent Sci. 2021 Jan;16(1):508-522. doi: 10.1016/j.jds.2020.06.019. Epub 2020 Jun 30. PMID 33384840
- [Background] Varela-Centelles P, Lopez-Cedrun JL, Fernandez-Sanroman J, Seoane-Romero JM, Santos de Melo N, Alvarez-Novoa P, Gomez I, Seoane J. Key points and time intervals for early diagnosis in symptomatic oral cancer: a systematic review. Int J Oral Maxillofac Surg. 2017 Jan;46(1):1-10. doi: 10.1016/j.ijom.2016.09.017. Epub 2016 Oct 15. PMID 27751768
- [Background] Seoane Leston JM, Aguado Santos A, Varela-Centelles PI, Vazquez Garcia J, Romero MA, Pias Villamor L. Oral mucosa: variations from normalcy, part I. Cutis. 2002 Feb;69(2):131-4. PMID 11871397
- [Background] Tanriver G, Soluk Tekkesin M, Ergen O. Automated Detection and Classification of Oral Lesions Using Deep Learning to Detect Oral Potentially Malignant Disorders. Cancers (Basel). 2021 Jun 2;13(11):2766. doi: 10.3390/cancers13112766. PMID 34199471